CLINICAL TRIAL: NCT06118528
Title: EAT: A Reliable Eating Assessment Technology for Free-living Individuals
Acronym: EAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU00215714; 1R01DK129843-01 (NIH)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Wearable Electronic Device
Keywords: Wearable; Electronic; Device; Behavior; Eat; Privacy; Camera; Obesity; Obfuscation; Filter; Cartoon; Blur; Raw; Edge; Burden; Wearer; Bystander; Monitor; BMI; Calories; Tool; Algorithm; RGB; Thermal; Data; Health; Chest
MeSH Terms: conditions — Behavior; Obesity | interventions — Airway Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blur Obfuscation (Experimental)
  Interventions: Device: Blur Obfuscation
- Edge Obfuscation (Experimental)
  Interventions: Device: Edge Obfuscation
- Cartoon Obfuscation (Experimental)
  Interventions: Device: Cartoon Obfuscation
- No Obfuscation (Raw) (Experimental)
  Interventions: Device: No Obfuscation (raw)

INTERVENTIONS:
Device: Blur Obfuscation — Blurring is applied to the RGB images.
  Arms: Blur Obfuscation
Device: Cartoon Obfuscation — Cartoonization is applied to the RGB images.
  Arms: Cartoon Obfuscation
Device: Edge Obfuscation — A black background and simple outlines of objects/people are applied to the RGB images.
  Arms: Edge Obfuscation
Device: No Obfuscation (raw) — No editing is performed on the RGB images.
  Arms: No Obfuscation (Raw)

SUMMARY:
This study utilizes a small, privacy-conscious wearable device intended to monitor human behaviors. The device is worn around the neck, capturing the wearer's head and upper torso within its field of view, and records color images without audio. Participants visit the lab for consent, device training and recording of several activities using the device. Participants will then take the device home and wear it during their normal schedules for four "active" weeks. During each active week, participants will wear the device, keep a log of all food and drink items consumed throughout the day and participate in unscheduled phone calls with a dietitian. A "washout" week occurs in between each active week in which participants do not need to complete any study tasks. Alongside the device, we have included three privacy filters (blur, edge, and avatar) capable of obscuring faces and objects seen in the device-captured images. All participants will be subject to unfiltered recording during their first week followed by a different filter each following active week in a random order. At the start of each active week, participants view an example of what their recorded images will look like that week (given the privacy filter). At the end of the seven weeks, participants will return the device and provide the lab with feedback on the design of the device and its privacy-preserving features.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 18.5
* Chicago metropolitan area resident
* Able to speak, read and write in English
* Has a valid phone number
* Owns a smartphone
* Has access to a computer

Exclusion Criteria:

* Pregnant or breastfeeding individuals
* Experienced significant weight loss/gain in the last three months (25 lbs or more)
* Diagnosed with or has a family history of genetic obesity syndromes (e.g., Prader-Willi, Bardet-Biedl, Cohen Syndrome)
* Member of household enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Daily wear time | 7 days

SECONDARY OUTCOMES:
Self-report acceptability | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT06118528/ICF_000.pdf